CLINICAL TRIAL: NCT04928794
Title: Dermatomal Spread of Paravertebral and Erector Spinae Plane Nerve Blocks as Compared by Thermal Imaging
Brief Title: Thermal-Imaging Comparison of Nerve Blocks for Bilateral Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Mary Billstrand, Associate Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-104 Billstrand
Record Dates: First submitted 2021-05-26; First posted 2021-06-16 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Conduction
Keywords: Paravertebral nerve block; Erector Spinae Plane block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral Nerve Block with 2 Techniques (Other)
  Interventions: Procedure: Erector Spinae Plane Block; Procedure: Paravertebral Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Regional anesthesia with injected local anesthetic solution, placed in space underlying erector spinae muscles
Procedure: Paravertebral Block — Regional anesthesia with injected local anesthetic solution, placed in space adjacent to vertebrae

SUMMARY:
This is a one-armed trial of two regional anesthesia (peripheral nerve block) techniques to provide postoperative analgesia after bilateral mastectomy. The two techniques are paravertebral block and erector spinae plane (ESP) block. Patients will serve as their own controls, with one block technique applied on one side of the body and the other technique contralaterally. Anatomical distribution of block effectiveness will be assessed with thermal imaging, and this distribution will be visually compared between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients having bilateral mastectomy surgery at University of New Mexico Outpatient Surgical and Imaging Services (OSIS) facility
* Age >18 years
* Consenting to regional anesthesia for postoperative pain control

Exclusion Criteria:

* Age <18 years
* Unable to consent
* Using anticoagulant medication or have a bleeding disorder
* Pregnancy
* Inability to speak English for consent process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Billstrand, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Outpatient Surgical and Imaging Services, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Anatomical side (Right vs Left)
Period: Overall Study
Arm/Group | Erector Spinae Plane Block | Paravertebral Block
Started | 8; 8 Anatomical side (Right vs Left) | 8; 8 Anatomical side (Right vs Left)
Completed | 8; 8 Anatomical side (Right vs Left) | 8; 8 Anatomical side (Right vs Left)
Not Completed | 0; 0 Anatomical side (Right vs Left) | 0; 0 Anatomical side (Right vs Left)

BASELINE CHARACTERISTICS:
Units Other Than Participants: Anatomical sides [Right vs Left]
Groups:
- Total: Total of all reporting groups
Arm/Group | Erector Spinae Plane Block | Paravertebral Block | Total
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (Anatomical sides [Right vs Left]) | 8 | 8 | 16
Age, Categorical [Count of Units; unit: Anatomical sides [Right vs Left]]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: Anatomical sides [Right vs Left]]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8
Superficial skin temperature [Mean (Standard Deviation); unit: degrees F] | 88.6 (1.7) | 88.6 (1.7) | 88.6 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Skin Temperature Increase From Baseline
Description: Thermography-measured increase in temperature of skin affected by nerve block
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: degrees C
Groups:
- Erector Spinae Plane Block Side: Side of body with Erector Spinae Plane Block
- Paravertebral Block Side: Side of body with Paravertebral Block
Arm/Group | Erector Spinae Plane Block Side | Paravertebral Block Side
Number analyzed (Participants) | 8 | 8
degrees C | 1.9 (0.8) | 2.3 (0.9)

2. Secondary Outcome: Average Skin Temperature
Description: Thermography-measured temperature of skin affected by nerve block
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Erector Spinae Plane Block Side | Paravertebral Block Side
Number analyzed (Participants) | 8 | 8
degrees C | 33.3 (0.9) | 33.7 (0.9)

ADVERSE EVENTS:
Time Frame: One day
Groups:
- Paravertebral Block: :Regional anesthesia with injected local anesthetic solution, placed in space adjacent to vertebrae
Arm/Group | Erector Spinae Plane Block | Paravertebral Block
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04928794/Prot_SAP_000.pdf